CLINICAL TRIAL: NCT05456204
Title: Efficacy and Safety of Refralon in Patients With Recurrent Atrial Fibrillation and Atrial Flutter After Catheter Ablation.
Brief Title: Refralon in Patients With Recurrence Paroxysmal and Persistent Forms of Atrial Fibrillation Who Underwent Catheter Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCBY-2021-0007-288
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Atrium; Fibrillation; Atrium; Flutter
Keywords: atrial fibrillation and flutter; paroxysmal and persistent atrial fibrillation and flutter; cardioversion AF; catheter radiofrequency ablation; Refralon; Niferidil; new antiarrhythmic drug; balloon cryoablation; reccurrence atrial fibrillation and flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refralone group (Other): Patients with recurrent AF/AFL after catheter interventions to restore SR will be cardioverted with refralon
  Interventions: Drug: Pharmacological cardioversion with Refralon

INTERVENTIONS:
Drug: Pharmacological cardioversion with Refralon — 1. the introduction of a 0.1% solution of refralon at a dose of 5 μg per 1 kg of body weight, diluted in 20 ml of saline intravenously for 2-3 minutes;
  2. in the absence of effect (SR recovery did not occur), after 15 minutes,repeated intravenous administration of a 0.1% solution of refralon at a dose of 5 μg per 1 kg of body weight (total dose of the drug 10 μg / kg of body weight);
  3. in the absence of effect (SR recovery did not occur),after 15 minutes, the next intravenous injection of a 0.1% solution of refralon at a dose of 10 μg per 1 kg of body weight (total dose of the drug 20 μg / kg of body weight);
  4. in the absence of effect (recovery of SR did not occur), after 15 minutes, repeated intravenous administration of a 0.1% solution of refralon at a dose of 10 μg per 1 kg of body weight. Thus, the maximum total dose of the drug will be 30 μg/kg of body weight.
  Other Names: Refralone

SUMMARY:
It is planned to evaluate the efficacy and safety of the class III antiarrhythmic drug refralon as a drug for pharmacological cardioversion in patients with recurrent atrial fibrillation (AF) and atrial flutter (AFL) after catheter ablation.

DETAILED DESCRIPTION:
Atrial fibrillation and atrial flutter are the most common arrhythmias among the adult population of the world, their share in the population is from 2 to 4% and continues to grow.

Modern highly effective methods of minimally invasive surgical treatment of these types of arrhythmia are currently catheter radiofrequency ablation and balloon cryoablation of the pulmonary veins. According to the CABANA study, catheter interventions reduce the risk of recurrent AF/AFL by 47%, significantly improving arrhythmia tolerance and improving the quality of life of patients.

An important problem is the recurrence of arrhythmia after the intervention, the frequency of recurrence of AF/AFL in the first 3 months after ablation (the so-called early recurrence) is 50-60%. In many patients, these recurrence are accompanied by severe clinical manifestations, which require pharmacological or electrical cardioversion.

In order to restore sinus rhythm, electrical cardioversion is most often used, the effectiveness of which is 90-92%.

An alternative to electrical cardioversion is pharmacological cardioversion, however, antiarrhythmic drugs used in wide clinical practice can restore sinus rhytm (SR) only in patients with recent AF paroxysms.

In 2014, a new Russian class III antiarrhythmic drug, Refralon, was registered. The effectiveness of the Refralon as a means of cardioversion in patients with persistent AF/AFL is 90%, in patients with paroxysmal AF/AFL - 95%.

At present, there is no information on the efficacy and safety of the use of refralon in patients with AF / AFL who underwent catheter ablation. The growing number of catheter ablation in the world dictates the to study new approaches to performing cardioversion in this cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

2. Patients with paroxysmal or persistent forms of AF/AFL and early (less than 90 days) or late (more than 90 days) arrhythmia recurrence after catheter radiofrequency ablation or balloon cryoablation of pulmonary veins.

3. Indications for SR recovery. 4. Consent of the patient.

Exclusion Criteria:

1. Arrhythmogenic effect of antiarrhythmic drugs III class in history;
2. Chronic kidney disease with a decrease in glomerular filtration rate less than 30 ml / min / 1.73 m2;
3. Chronic heart failure (functional class IV);
4. Acute coronary syndrome;
5. Bronchial asthma of an uncontrolled course and / or severe respiratory failure.
6. The need for the use of drugs that increase the duration of the QT interval drugs without the possibility of withdrawal
7. Atrioventricular blockade of 2-3 degrees (with the exception of patients with an implanted pacemaker);
8. Dysfunction of the sinoatrial node (with the exception of patients with an implanted pacemaker);
9. Bradysystolic atrial fibrillation (heart rate <50 beats/min);
10. Duration of the QT interval >440 ms;
11. Hemodynamic instability requiring emergency cardioversion;
12. Contraindications to anticoagulant therapy;
13. Thyrotoxicosis or decompensated hypothyroidism;
14. Uncorrected electrolyte disturbances at the time of cardioversion (potassium level less than 3.5 mmol/l);
15. Pregnancy and breastfeeding period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Restoration of sinus rhythm | 24 hour
  Restoration of SR within 24 hours from the moment of administration of the first dose of refraloRestoration of SR within 24 hours from the moment of administration of the first dose of refralon
Preservation of SR | 24 hours
  Preservation of SR 24 hours after the first dose of refralon.
Ventricular arrhythmogenic effect | 24 hours
  Registration of sustained and nonsustained (3 or more QRS) ventricular tachycardia or ventricular fibrillation after administration of drug
Increased QT interval (more than 500 ms) | 24 hours
  The number of patients who have an increase in the QT interval (more than 500 ms) and the time during which the duration of the QT interval exceeded 500 ms.

SECONDARY OUTCOMES:
Restoration of sinus rhythm within 6 hours | 6 hours
  Restoration of SR within 6 hours from the moment of administration of the first dose of refralon
Number of patients recovering SR after minimal doses | 24 hours
  Number of patients who recovered SR after minimal doses of refralon (5-10 μg/kg)
Reccurence after SR recovery | 24 hours
  Absence of sustained (lasting more than 30 seconds) recurrences of AF/AFL within 24 hours after successful recovery of SR with refralon
Bradyarrhythmias (pauses and bradycardia) | 24 hours
  Decrease in heart rate to less than 50bpm after administration of drug (refralon/amiodarone) during AF or after restoration of SR - the minimum heart rate, the duration of the maximum recorded pause and the time during which the heart rate was less than 50bpm will be recorded
Pauses more than 5 seconds | 24 hours
  The presence of pauses for more than 5 seconds at the time of SR recovery or against the background of persistent AF/AT.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution NATIONAL MEDICAL RESEARCH CENTRE OF CARDIOLOGY NAMED AFTER ACADEMICIAN E.I.CHAZOV. of the Ministry of Health of the Russian Federation, Moscow, Russia